CLINICAL TRIAL: NCT02784769
Title: Role of Molecular Aging of Matrix Proteins of the Vessel Wall in the Aneurysm Pathology
Brief Title: Matrix Aging and Aneurysm
Acronym: VIMANE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO14056
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2018-04

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

ARMS (2):
- aneurysm diameter of below 75 mm (Experimental)
  Interventions: Other: measurement of skin autofluorescence; Other: skin biopsy collection
- aneurysm diameter above 75 mm (Experimental)
  Interventions: Other: measurement of skin autofluorescence; Other: skin biopsy collection

INTERVENTIONS:
Other: measurement of skin autofluorescence
Other: skin biopsy collection

SUMMARY:
During their biological life, proteins undergo molecular aging due to many non-enzymatic post-translational modifications that alter their structural and functional properties. These reactions concern all proteins but especially tissue proteins (whose half-life in the organism can be several decades) and lead to the formation of complex products called PTMDPs ("post-translational modification derived products"). Molecular aging is responsible for the alteration of protein properties which may cause changes in mechanical properties of tissues during aging and pathologies. However, the involvement of these processes in vivo remains unclear, particularly in the aneurysmal pathology. So, the aim of this study is to determine whether the molecular aging of matrix proteins within the vessel wall may participate in the development of aortic aneurysm.

DETAILED DESCRIPTION:
The investigators hypothesized that the molecular aging of matrix proteins may participate in the formation of aortic aneurysm. Indeed, it is well known that the aneurysm wall is subjected to important structural changes including variations in extracellular matrix composition. However, few studies have looked for a link between the molecular aging of matrix proteins and the formation of aneurysm. So, the aim of this study is to understand the role of protein molecular aging in this context.

For that purpose, several approaches will be used to reach this aim: (1) To evaluate the degree of modification of matrix components at the aneurysmal wall by biological and histological studies (concentrations of PTMDPs (homocitrulline, carboxymethyllysine, pentosidine and MG-H1) and expression of RAGE) ; (2) To determine if there is a link between tissue concentrations of PTMDPs and the severity of the aneurysmal pathology ; (3) To compare concentrations of PTMDPs obtained at the aneurysmal wall with those obtained in skin and serum ; (4) To establish a link between concentrations of PTMDPs (in serum, skin and vascular wall), fragmentation of elastin and different haematological parameters potentially involved in the development of the pathology aneurysmal.

Design of the study: single-center cross-sectional study. Population: 40 patients with aneurysm of the infra-renal abdominal aorta requiring surgical treatment by open surgery. Patients will be divided into 2 groups based on the size of the aneurysm (Group 1: 20 patients with aneurysm diameter of below 75 mm; Group 2: 20 patients with aneurysm diameter above 75 mm; patients a ruptured aneurysm can be included in both groups).

Investigation scheme: after obtaining the inform consent of the patient, several samples or investigations will be done: blood (PTMDPs and hematological paramaters), measurement of skin autofluorescence (AGE-Reader), skin biopsy collection (2 to 3 mm wide and a few centimeters during the laparotomy), a biopsy of both aneurysmal and not aneurysmal aortic wall (from the abdominal aorta fragment usually resected part of the surgery and therefore being surgical waste) and collection of intra-aneurysmal and peri-thrombotic liquid (if available).

Statistical analyses: (1) Description of data using mean and standard deviation for quantitative variables and percentage for qualitative variables. (2) Comparison of PTMDP concentrations between patient groups and between tissue locations (healthy or aortic aneurysms) using the Mann-Whitney test. (3) Search for links between concentrations of tissue PTMDPs, serum, skin autofluorescence, and hematologic markers using the Spearman correlation tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aneurysm of the infrarenal abdominal aorta requiring surgical care by open surgery.
* Patients older than 18 years.
* Patients who agreed to participate in the study.

Exclusion Criteria:

* Patients with aneurysm of the abdominal infrarenal aorta due to trauma or infection.
* Patients who have already received surgery for an aneurysm of abdominal aorta.
* Patients who are protected by law.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11-22 (Actual); Study Completion 2016-11-22 (Actual)

PRIMARY OUTCOMES:
blood collection | at the same time of surgery
measurement of skin autofluorescence with AGE-reader (Diagnoptics®) | at the same time of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Background] Doue M, Marques G, Okwieka A, Gorisse L, Pietrement C, Gillery P, Jaisson S. Accumulation of Carbamylation-Derived Products in Aneurysmal Aorta. J Vasc Res. 2024;61(2):51-58. doi: 10.1159/000534613. Epub 2024 Jan 19. PMID 38246153